CLINICAL TRIAL: NCT02773706
Title: Detecting and Evaluating Childhood and Anxiety and Depression Effectively in Subspecialties
Acronym: DECADES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, William E. Bennett, Jr., Assistant Professor of Pediatrics, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DECADES
Record Dates: First submitted 2015-06-19; First posted 2016-05-16 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Subspecialty Care (Experimental): Once a subject is screened positive for anxiety or depression, the subspecialty provider is informed of the positive screen, and left to manage or refer the condition as per usual care by that provider.
  Intervention: Depression / anxiety screen + clinician informed.
  Interventions: Other: Notification of Subspecialist
- Integrated Psychology Care (Active Comparator): Once a subject is screened positive for anxiety or depression, an automated psychology referral occurs, in addition to any intervention determined by the subspecialty provider.
  Intervention: Depression / anxiety screen + clinician informed + automated psychologist visit.
  Interventions: Other: Automated Psychology Services

INTERVENTIONS:
Other: Automated Psychology Services — The automated screening tool determines a positive or negative screen, then informs the clinician, and also automates a psychology visit.
  Arms: Integrated Psychology Care
Other: Notification of Subspecialist — The automated screening tool determines a positive or negative screen, then informs the clinician.
  Arms: Usual Subspecialty Care

SUMMARY:
The DECADES trial seeks to determine the comparative effectiveness of specialist-centered management of anxiety and depression vs. an imbedded and automated psychology referral for all subjects who screen positive for anxiety or depression.

DETAILED DESCRIPTION:
SPECIFIC AIMS: Mental Health and Quality of Life in Children with Gastrointestinal Disorders Depression and anxiety are two of the most common and dangerous disorders in childhood and adolescence. Currently, a large proportion of children with these disorders remain unrecognized or untreated resulting in considerable morbidity and mortality. The rates of depression and anxiety are significantly higher in children with chronic illnesses, including gastrointestinal disorders, than in the general population. Furthermore, children with depression or anxiety are far more likely to have somatic complaints, and have greater utilization of subspecialty care, especially in gastroenterology. Functional gastrointestinal disorders such as irritable bowel syndrome, chronic recurrent abdominal pain, and functional dyspepsia frequently have comorbid anxiety or depression.

Efforts to recognize and treat mental health problems in children with chronic medical illness, such as gastrointestinal disorders, have been shown to improve adherence to therapy, as well as other clinical outcomes. More importantly, improving such mental health problems might go far to addressing the outcomes patients care about most with respect to their gastroenterological disease. Unfortunately, mental health resources are often difficult for families to access, even when these disorders are recognized.

Validated screening tools exist to screen for anxiety and depression in children and adolescents, including the Screen for Childhood Anxiety Related Emotional Disorders (SCARED) and the Patient Health Questionnaire (PHQ-9). Despite the established importance of depression and anxiety in the gastrointestinal health of children and adolescents, few data exist describing the treatment of anxiety and depression by pediatric gastroenterologists. Furthermore, little is known about how families or patients view the subspecialty office as the setting to detect or care for mental illness. Additionally, if anxiety and depression are identified by the gastroenterologist, many practitioners find either they have limited training and expertise in the management of adolescent mental health disorders, or they encounter barriers to referral to a mental health specialist, especially in children with public insurance.

Therefore, the specific aims of this research project are to:

Aim 1: Determine family and patient attitudes towards tools to screen for mental illness in a pediatric subspecialty office utilizing structured interviews.

Sub Aim 1a: Determine patient and family attitudes toward anxiety and depression screening in a subspecialty office.

Sub Aim 1b: Determine outcomes of importance to patients and families related to anxiety and depression in a pediatric subspecialty office.

Aim 2: Develop an integrated approach that accounts for family and patient preferences as determined in Aim 1, to deliver anxiety and depression screening instruments to new and established patients in a pediatric gastroenterology clinic.

Aim 3: Perform a pre-post comparative effectiveness trial comparing screening in a pediatric gastroenterological clinic with notification of the physician to screening in a pediatric gastroenterological clinic with the addition of a psychologist, with respect to the patient-centered outcomes identified in Aim 1.

Completion of these aims will allow the investigators to develop an integrated process to screen for depression and anxiety in a high-risk population. Furthermore, the knowledge gained from piloting depression and anxiety screening will help the investigators to determine attitudes towards this approach in the pediatric subspecialty setting, which will maximize outcomes from the visit that are important to patients and their families.

The investigators hypothesize that a combined approach that screens for depression and anxiety within the gastroenterology clinic and also provides for access to a psychologist who is integrated with the clinic will lead to superior clinical and patient-centered outcomes. However the investigators may find that screening patients and then alerting the gastroenterology provider may be sufficient to recognize and treat mental health disorders effectively. Comparing the effectiveness of these two strategies is therefore important and is the overall focus of this proposal.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen at the pediatric GI office who are screened for anxiety and depression as part of usual care.

Exclusion Criteria:

* Patients over the age of 18 or under the age of 10.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Quality of life (baseline) | Baseline
  Baseline quality of life measurement will be determined using the PedsQL instrument. Both the general PedsQL instrument and the PedsQL gastroenterology symptom index will be used for baseline and followup measures.
  PedsQL Minimum score: 0 (Worse outcome) PedsQL Maximum score: 100 (Better outcome)
Quality of life (followup) | Within 6 months
  Baseline quality of life measurement will be determined using the PedsQL instrument. Both the general PedsQL instrument and the PedsQL gastroenterology symptom index will be used for baseline and followup measures.
  PedsQL Minimum score: 0 (Worse outcome) PedsQL Maximum score: 100 (Better outcome)

SECONDARY OUTCOMES:
Utilization of endoscopy | Within 6 months
  The investigators will compare the use of endoscopy, radiologic testing, laboratory testing, emergency department utilization, and repeat gastroenterology outpatient visits. Frequency of each of these will be compared between control and intervention arms.
Utilization of radiologic testing | 6 months
  The electronic medical record will be queried by the RA and the total number of radiologic tests ordered over 6 months will be computed.
Utilization of laboratory testing | 6 months
  The electronic medical record will be queried by the RA and the total number of laboratory tests ordered over 6 months will be computed.
Utilization of emergency department visits | 6 months
  The electronic medical record will be queried by the RA and the total number of emergency department visits over 6 months will be computed.
Utilization of outpatient gastroenterology | 6 months
  The electronic medical record will be queried by the RA and the total number of outpatient gastroenterology visits over 6 months will be computed.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health North Hospital, Carmel, Indiana, United States

IPD SHARING:
Plan to Share IPD: No